

Version 3: 23.04.2020 IRAS 250408







## **Consent Form**

The effects of a fasted versus fed remote walking-based training Title of Project: programme on glycaemic control in overweight individuals

| Name | of Researchers: | Ms Jennifer Barrett, D<br>Anton Wagenmakers | Or Juliette Strauss, Dr Daniel Cuthbertson, P<br>, Dr Sam Shepherd | rofessor |
|---|---|---|---|---|
| | | | Please in | itial all boxes |
| 1. | I confirm that I have read and understand the information sheet dated 23.04.20 (version 3) for the above study. I have had the opportunity to consider the information, ask questions and have had these answered satisfactorily. | | | |
| 2. | I understand that my participation is voluntary and that I am free to withdraw at any time without giving any reason, without my medical care or legal rights being affected. I also understand that if I withdraw from the study the data already collected will be retained, unless I request for it to be removed within I2 weeks of the first visit. | | | |
| 3. | I understand that the sponsor and regulatory body may require access to research records for monitoring purposes. | | | |
| 4. | I confirm that the research team will contact my GP to inform them of my involvement in the study. | | | |
| 5. | I agree to take part in the above study. | | | |
| _ | Name of participant | Date | Signature | |
| | Name of person taking<br>consent | Date | Signature | |

When completed: I copy for participants, I for research site file, I (original) to be kept in notes.